CLINICAL TRIAL: NCT05314543
Title: Description and Determinants of the Power-speed-endurance Profile (PVE) in Cycling and Rowing to Optimize the Performance of the French Athletes at the Paris Olympics 2024
Brief Title: Power-speed-endurance Profile (Cycling/Rowing) : Optimize Performance of the French Athletes at the Paris Olympics 2024
Acronym: THPCA2024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21CH145; 2021-A02341-40 (Other: ANSM)
Record Dates: First submitted 2022-02-02; First posted 2022-04-06 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers; Performance
Keywords: Biomechanics; Track cyclists and rowers; Energetics; Muscle; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: This is a prospective multi-center exploratory pilot study of physiology study on athletes, track cyclists or rowers national to international level competitors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Track cyclists and rowers (males and females) (Experimental): All female and male rowing and track cycling athletes at the national or international national or international level, registered in a selection process and likely to represent France at the likely to represent France at the 2024 Olympics will be asked to take part to take part in this study.
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — Subjects will be subjected to mild hypoxia simulating an altitude of 1750 m (normobaric hypoxia). Hypoxia decreases oxygen supply to tissue and limit exercise capacity. For this, the subjects will inhale a gas mixture depleted in oxygen (enriched in nitrogen). The barometric pressure at 1500 m being 621 mmHg, PIO2 at this altitude (PIO2 = (621 - 47) x 21%) is 120.5 mmHg. For sea level altitude where the barometric pressure is 760 mmHg, the hypoxic gas mixture should contain (x = 120.5 / (760 - 47)) 16.8% O2. Thus, by inhaling a gas mixture that is oxygen-depleted from 21 to 16.8%, subjects (will simulate the altitude of 1750 and) will experience the equivalent of a 20% reduction in oxygen supply.

SUMMARY:
As part of the preparation at the Paris 2024 Olympic Games, the French rowing and cycling federations and a consortium of researchers met to reach an ultimate goal: to increase the number of medals in these two disciplines for Paris 2024 Olympics.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the maximum capacity of power production of athletes by describing their power-endurance profile and the physiological factors underlying this maximum power generation capacity. These assessments will guide coaches and athletes for:

1. the best use of athletes' physical abilities (for race strategy, cycling gear ratio or rowing levers)
2. adaptation of training program to improve the maximum capacity of power production of the athletes, in order to increase the number of medals at the Paris Olympics 2024.

ELIGIBILITY:
Inclusion Criteria:

* experienced, well-trained (national to international level) rowers and cyclists
* written consent

Exclusion Criteria:

* taking medications interfering with measured parameters
* contraindication to competitive sport practice
* currently participating in an other structured exercise program
* muscular, bone or joint injuries
* neurologic disease
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum force produced at zero speed in a fatigue-free condition | Month : 3
  F0i measurement
Speed in a fatigue-free condition | Month : 3
  V0i measurement
Maximum force produced at zero speed at the end of the 3 min. | Month : 3
  F0e measurement
Speed up produced at the end of the 3 min. | Month : 3
  V0e measurement

SECONDARY OUTCOMES:
Maximal oxygen uptake (VO2max) | At inclusion
  Cardiac stress test
Maximal Ventilation (VEmax) | At inclusion
  Cardiac stress test
Cardiac output (QCmax) | At inclusion
  Cardiac stress test
Maximal cardiac frequency (fcmax) | At inclusion
  Cardiac stress test
Fibre type determination | Month : 2
  Muscle biopsy of the vastus lateralis
Microvasculature analysis | Month : 2
  Muscle biopsy of the vastus lateralis
Muscle enzyme activity (Phosphofructokinase (PFK), lactate dehydrogenase (LDH), citrate synthase (CS) et cyclo-oxygenase (COx)) | Month : 2
  Muscle biopsy of the vastus lateralis
Maximal voluntary force (N) | Month : 9
  Comparison before and after exercise
Rate of force development | Month : 9
  Comparison of force development
Evoked forces (N) | Month : 9
  Ratio of evoked force at low and high frequencies
Maximum force produced at zero speed in a fatigue-free condition after bicarbonate ingestion | Month : 3
  F0i measurement
Speed in a fatigue-free condition after bicarbonate ingestion | Month : 3
  V0i measurement
Maximum force produced at zero speed at the end of the 3 min after bicarbonate ingestion | Month : 3
  F0e measurement
Speed up produced at the end of the 3 min after bicarbonate ingestion | Month : 3
  V0i measurement
Maximal oxygen uptake (VO2max) after bicarbonate ingestion | At inclusion
  Cardiac stress test
Maximal Ventilation (VEmax) after bicarbonate ingestion | At inclusion
  Cardiac stress test
Cardiac output (QCmax) after bicarbonate ingestion | At inclusion
  Cardiac stress test
Maximal cardiac frequency (fcmax) after bicarbonate ingestion | At inclusion
  Cardiac stress test
Fibre type determination after bicarbonate ingestion | Month : 2
  Muscle biopsy of the vastus lateralis
Microvasculature analysis after bicarbonate ingestion | Month : 2
  Muscle biopsy of the vastus lateralis
Muscle enzyme activity (Phosphofructokinase (PFK), lactate dehydrogenase (LDH), citrate synthase (CS) et cyclo-oxygenase (COx)) after bicarbonate ingestion | Month : 2
  Muscle biopsy of the vastus lateralis
Maximal voluntary force (N) after bicarbonate ingestion | Month : 9
  Comparison before and after exercise
Rate of force development after bicarbonate ingestion | Month : 9
  Comparison of force development
Evoked forces (N) after bicarbonate ingestion | Month : 9
  Ratio of evoked force at low and high frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, PhD, Principal Investigator — CHU SAINT-ETIENNE; Laurent MESSONNIER, PhD, Study Director — Université Savoie Mont Blanc, CHAMBERY
Locations (3):
- France (3):
  - CEPART, Le Bourget-du-Lac
  - Chu Nantes, Nantes
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No